CLINICAL TRIAL: NCT06258525
Title: A Phase II, Open-Label Trial of S-Adenosylmethionine (SAMe) in Prevention of Oxaliplatin Associated Liver Injury
Brief Title: SAMe in Prevention of Oxaliplatin-associated Liver Injury
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Jarrow Formulas Inc (Industry)
Responsible Party: Principal Investigator, Alexandra Gangi, MD, Sponsor-Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2022-11-Gangi-SAMe
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Liver Metastases; Liver Metastasis Colon Cancer; Liver Injury; Sinusoidal Obstruction Syndrome; 5-Fluorouracil Toxicity; Liver Toxicity, Chemically-Induced
Keywords: S-adenosylmethionine; Oxaliplatin; Stage IV colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Hepatic Veno-Occlusive Disease; Chemical and Drug Induced Liver Injury | interventions — S-Adenosylmethionine; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Radiation: Standard of care oxaliplatin-based chemotherapy; Dietary Supplement: S-adenosylmethionine (SAMe) supplement; Procedure: Surgery

INTERVENTIONS:
Radiation: Standard of care oxaliplatin-based chemotherapy — mFOLFOX6 or CAPOX
Dietary Supplement: S-adenosylmethionine (SAMe) supplement — (400 mg tablet): 2 tablets taken orally AM and 1 tablet PM daily (total 1,200 mg daily) prior to surgical resection
Procedure: Surgery — At 1-Month

SUMMARY:
This is an open-label, phase II study that may provide evidence that taking S-adenosylmethionine (SAMe) supplementation prevents oxaliplatin, a type of chemotherapy drug, associated liver toxicity in patients with resectable colorectal liver metastases. Resectable means that it is able to removed with surgery. Patients will take two SAMe tablets in the morning and one tablet in the evening for 3-6 months (about 6-8 cycles of chemotherapy) in addition to oxaliplatin based chemotherapy followed by surgical removal of the colorectal liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV patients with resectable liver predominant metastatic colorectal cancer (new diagnosis or recurrent) referred to Cedars Sinai Medical Center for oxaliplatin based systemic therapy.
* Age ≥ 18 years.
* Patients who are planning to undergo liver resection following oxaliplatin based chemotherapy treatment.
* ECOG Performance Status 0-2 or Karnofsky Performance Status (KPS) ≥ 60%.
* Demonstrate adequate organ and marrow function (within 28 days of study treatment initiation)
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 14 days prior to receiving the first dose of study medication for eligibility verification purposes. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use adequate methods of birth control (hormonal or barrier method of birth control) or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of therapy through 120 days after the last dose of therapy.
* Subjects taking vitamin E ≥800 IU/day must be on a stable dose defined as:

  1. No changes in prescribed dose within 180 days of the screening visit and
  2. No new vitamin E-containing medications within 180 days of the screening visit or
  3. Discontinuation of vitamin E ≥800 IU/day for at least 180 days prior to the screening visit.
* Subjects taking anti-diabetic medications must be on a stable dose for at least 90 days prior to the date of the screening visit.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* No other anti-cancer therapy (chemotherapy, hormonal therapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) or investigational agent may be used from 28 days prior to registration and until the end-of-study visit.
* Has previously received chemotherapy for metastatic disease (neoadjuvant or adjuvant therapy is allowed as long as treatment was completed ≥6 months prior to recurrence).
* Has pre-existing grade ≥ 3 neuropathy precluding use of oxaliplatin.
* Has known additional malignancy that is progressing or requires active treatment.
* Has a known hypersensitivity to any of the study supplement/drugs (SAMe, oxaliplatin, flourouacil, folinic acid and capecitabine).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has any gastrointestinal disorder (e.g., bowel obstruction) or neurologic condition (e.g., oropharyngeal dysphagia) that may result in impairment of oral intake, inability to swallow the oral supplement, and/or impairment of absorption of study drug in the opinion of the treating investigator.
* Has previous clinical diagnosis of cirrhosis, has had known history of Hep A/B/C or nonalcoholic fatty liver disease (NAFLD), liver transplantation, or any other cause for decompensated liver disease.
* Known human immunodeficiency virus (HIV) infection.
* Any of the following within 6 months prior to the screening visit: unstable cardiovascular disease, myocardial infarction, coronary artery bypass surgery, coronary angioplasty, transient ischemic attack, or cerebrovascular accident.
* Any other condition that, in the investigator's opinion, would impede competence or compliance or delay completion of the study.
* History of Parkinson's disease or bipolar disorder.

Patients taking the following prohibited medications:

* Olanzapine
* MAO inhibiters, including:

  * Isocarboxazid
  * Linezolid
  * Methylene blue injection
  * Phenelzine
  * Rasagiline
  * Selegiline
  * Tranylcypromine
  * Any other MAO inhibitors The above prohibited medications cannot be taken -14 days prior to Day 0 and during study treatment.. Patients currently on or plan to be prescribed anti-psychotic medications not listed above may be excluded at the discretion of the Investigator. - Active infection as evidenced by positive urine culture, blood culture, or pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of SAMe in preventing oxaliplatin associated liver injury as determined by lack of injury on histopathologic analysis in patients with liver only stage IV colorectal cancer. | 8 months
  To identify the effect of SAMe in preventing oxaliplatin associated liver injury as determined by lack of injury on histopathologic analysis in patients with liver only stage IV colorectal cancer. Improvement in liver injury will be measured by the degree/histopathologic grade of liver injury utilizing the Combined Vascular Injury (CVI) Score in non-cancerous liver tissue post therapy compared to historical controls. CVI score will evaluate and grade sinusoidal dilation, small vessel loss/obliteration, focal hepatocyte plate disruption, parenchymal extinction lesions, nodular regenerative hyperplasia, peliosis, and veno-occlusive like changes. Rate of sinusoidal obstruction syndrome (SOS), as measured by CVI Score, ranging from 0-13. A CVI score of 3 or more indicates SOS. Compared to historical controls.

SECONDARY OUTCOMES:
To Estimate the Objective Response Rate (ORR) of SAMe when taken with oxaliplatin based chemotherapy. | 8 months
  To evaluate the efficacy of SAMe during oxaliplatin based therapy in stage IV liver-only colorectal cancer, Objective Response Rate (ORR) will be measured by the proportion of patients with confirmed complete response (CR) or partial response (PR) per RECIST 1.1. ORR will be assessed from screening until EOT.
To evaluate changes in average estimated blood loss (EBL) in patients undergoing liver resection as compared to historical controls. | 8 months
  Calculate surgical EBL in all patients undergoing resection
To evaluate length of hospital stay (LOS) in patients undergoing liver resection as compared to historical controls. | 8 months
  Length of hospital stay (LOS) to historical controls, the following will be conducted:
  ii. Calculate hospital LOS in all patients undergoing resection iii. Account for 30-day readmission
To examine if SAMe can decrease treatment-delays in oxaliplatin-based chemotherapy. | 8 months
  Incidence of oxaliplatin treatment delays will be evaluated by recording the following: If treatment delay occurred and time point/duration of treatment delay
To examine if SAMe can decrease dose-reductions in oxaliplatin-based chemotherapy. | 8 months
  Incidence of oxaliplatin dose reduction will be evaluated by recording the following: If dose reduction occurred and time point of occurrence
To evaluate safety and tolerability of SAMe in combination with SOC oxaliplatin based systemic therapy. | 8 months
  Safety and tolerability of the combination will be evaluated by determining the proportion of patients with treatment-related adverse events of all grades as graded per CTCAE v.5, from first dose of study drug until 30 days post last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Gangi, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center at SOCC, Los Angeles, California
  - Cedars-Sinai Medical Center Beverly Hills, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No